CLINICAL TRIAL: NCT04532658
Title: Understanding the Influence of Human and Organizational Factors on Surgeon Performance to Enhance Patient Outcomes: Experimental Evaluation of a Customized Coaching Program
Brief Title: Evaluation of Coaching Impact on Surgical Outcomes
Acronym: TopSurgeons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TOPSURGEONS_2020
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Surgeons randomly assigned to the intervention arm
  Interventions: Behavioral: Coaching program
- Control arm (No Intervention): Surgeons randomly assigned to the control arm

INTERVENTIONS:
Behavioral: Coaching program — * Charting system for outcomes feedback
  * Profiling of individual surgeon
  * Modules of improvement
  Arms: Intervention arm

SUMMARY:
This two arms parallel cluster-randomized trial will evaluate the impact of a customized coaching program for surgeons on the occurrence of patient major adverse events. Trends in surgical outcomes before and after the intervention will be compared between surgeons randomly assigned to the coaching program against non-exposed surgeons.

ELIGIBILITY:
Inclusion Criteria:

* All adults needing a surgery who are operated by one of the participating surgeons

Exclusion Criteria:

* Age < 18 years old
* Absence of surgical procedure
* Palliative care
* Organ transplantation
* Refusal for personal data sharing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20791 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of major adverse event | During surgery or within 30 days after the operation
Occurrence of death | During surgery or within 30 days after the operation
Occurrence of unplanned stay in critical/intensive care unit | Within 30 days after the operation
Occurrence of unplanned reoperation | Within 30 days after the operation
Occurrence of intraoperative and postoperative complications | During surgery or within 30 days after the operation
: Occurrence of avoidable hospital readmission for complication | Within 30 days after the operation
Operative time | From skin incision to wound closure
Length of stay | From hospital admission to discharge, within 30 days after operation
Hospitalization costs | Within 30 days after the operation
Surgeon well-being | Throughout the study, Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://topsurgeons.univ-lyon1.fr